CLINICAL TRIAL: NCT01760421
Title: The Effect of Hydroxychloroquine Treatment in Hashimoto's Thyroiditis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201108006MB
Record Dates: First submitted 2011-10-20; First posted 2013-01-04 (Estimated); Last update posted 2014-04-23 (Estimated); Status verified 2014-04

CONDITIONS: Hashimoto Thyroiditis
MeSH Terms: conditions — Hashimoto Disease | interventions — Hydroxychloroquine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Hydroxychloroquine (Experimental): Receive treatment with hydroxychloroquine
  Interventions: Drug: Hydroxychloroquine

INTERVENTIONS:
Drug: Hydroxychloroquine — Hydroxychloroquine (200mg/tab) 1 tab twice daily orally for 6 months
  Other Names: Plaquenil

SUMMARY:
Hashimoto's thyroiditis is an autoimmune thyroid disease, which induced chronic inflammation of thyroid gland and destroys thyroid tissue.

Hydroxychloroquine is used as disease modifying anti-rheumatic drug (DMARD) for treatment of several autoimmune diseases, such as systemic lupus erythematosus (SLE), rheumatoid arthritis(RA) for more than one century.

The purpose of this study is to evaluate whether hydroxychloroquine is effective in treatment of Hashimoto's thyroiditis.

DETAILED DESCRIPTION:
Hashimoto's thyroiditis is an autoimmune thyroid disease, and when the disease progresses, thyroid function finally declined to hypothyroidism.

There was no medical treatment recommended for patients with Hashimoto's thyroiditis, but currently at euthyroid state. Levothyroxine replacement therapy starts if patients become hypothyroid state.

Hashimoto's thyroiditis is a T-cell mediated autoimmune thyroid disease. The major auto-antigens include thyroid peroxidase (TPO) and thyroglobulin. Anti-TPO antibodies induce antibody-dependent cell-mediated cytotoxicity (ADCC) and cause destruction of thyroid tissues.

Antimalarial agents like hydroxychloroquine have several pharmacologic effects which may be involved in the treatment of rheumatic diseases, but the role of each is not known. These include interaction with sulphydryl groups, interference with enzyme activity (including phospholipase, nicotinamide adenine dinucleotide hydrogen-cytochrome C reductase, cholinesterase, proteases and hydrolases), DNA binding, stabilisation of lysosome membranes, inhibition of prostaglandin formation, inhibition of polymorphonuclear cell chemotaxis and phagocytosis.

This study is to investigate the treatment effect of hydroxychloroquine on autoantibodies and disease progression of Hashimoto's thyroiditis.

ELIGIBILITY:
Inclusion Criteria:

* Hashimoto's thyroiditis
* Euthyroid state (free T4 and thyroid-stimulating hormone level within normal limit)
* Never receive immunomodulators or immunosuppressants

Exclusion Criteria:

* Planned pregnant or already pregnant women
* Renal insufficiency
* Hepatic insufficiency
* Anemia
* Agranulocytosis
* Thrombocytopenia
* Glucose-6-phosphate dehydrogenase deficiency
* Porphyria cutaneous tarda
* Allergy to 4-aminoquinolone

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2011-10; Primary Completion 2012-12 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Anti-TPO antibody | 6th month after medical treatment
  Check anti-TPO antibody 6 months after medical treatment as inflammatory marker
Anti-thyroglobulin antibody | 6 months after medical treatment
  Check serum anti-thyroglobulin antibody 6 months after medical treatment as inflammatory status

SECONDARY OUTCOMES:
Elasticity of thyroid gland | 6 months after medical treatment
  Measure the elasticity of the thyroid gland by elastography as the infiltrative degree of the thyroid
Thyroid function | 6 months after medical treatment
  Measure serum free T4 and thyroid-stimulating hormone level 6 months after treatment
Inflammatory cytokines | 6 months after treatment
  Measure plasma cytokines including interleukin-1, interleukin-6, tumor necrosis factor-alpha, 6 months after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Tien-Shung Huang, Ph.D., Study Chair — Department of Internal Medicine, National Taiwan University Hospital, Taipei, Taiwan
Locations (1):
- Department of Internal Medicine, National Taiwan University Hospital, Taipei, Taiwan, Taiwan